CLINICAL TRIAL: NCT03815318
Title: A Multicenter, Open, Single Arm Evaluation of the Efficacy, Safety and Pharmacokinetics of Recombinant Human Coagulation FVIII (SCT800) in Prophylaxis Therapy on Patients With Severe Hemophilia A Who Had Previously Treated With FVIII.
Brief Title: Evaluation of SCT800 in Prophylaxis Therapy on Previous Treated Patients With Severe Hemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other); Parexel (Industry); Q2 Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SCT800-A 302
Record Dates: First submitted 2019-01-17; First posted 2019-01-24 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recombinant Human Coagulation FVIII (Experimental): Participant receivedSCT800 for prophylaxis with 25 - 50 IU/kg injection once every other day or three times per week for 6 months.
  Interventions: Drug: Recombinant Human Coagulation FVIII

INTERVENTIONS:
Drug: Recombinant Human Coagulation FVIII — Participant received SCT800 for prophylaxis with 25 - 50 IU/kg injection once every other day or three times per week for 6 months.
  Other Names: SCT800

SUMMARY:
This study is a multi-center, open-label, single-arm trial to evaluate the efficacy,safety and pharmacokinetics of SCT800 in regular prophylaxis and perioperative treatment in patients (≥12 years old) with severe hemophilia A who have been previously treated with coagulation factor VIII(FVIII:C) . This study includes two phases: the screening period and prophylaxis period.Prophylaxis with 25 - 50 IU/kg of SCT800 shall be administered once every other day or three times per week starting from V1 and prophylaxis with SCT800 shall continue for 24 consecutive weeks.

DETAILED DESCRIPTION:
After subjects pass screening, prophylaxis with 25 - 50 IU/kg of SCT800 shall be administered once every other day or three times per week for 6 months. Subjects shall receive FVIII intravenous injection treatment at the study site or at home. During the study prophylaxis treatment period, subjects should return for visit every four weeks, namely for Visit (V) 2 (4 weeks ± 4 days), Visit 3 (8 weeks ± 4 days), Visit 4 (12 weeks ± 4 days), Visit 5 (16 weeks ± 7 days), Visit 6 (20 weeks ± 7 days), Visit 7 (24 weeks ± 7 days) and end-of-treatment (EOT) visit (+ 14 days). Of which, blood collection shall be carried out during the screening period and in V1, V2, V4, V7 and the EOT visit for FVIII inhibitor assay; blood collection shall be carried out before and after the completion of SCT800 infusion in V1, V4 and V7 for incremental in-vivo recovery (IVR) assay.

FVIII:C activity shall be monitored before injection and 15minutes(min), 30min, 1h, 3h, 6h, 9h, 12h, 24hours(h), 28h, 32h and 48h after injection at V1 and V7. Then pharmacokinetics parameters (incremental in-vivo recovery, t1/2 etc.) of SCT800 shall be calculated and evaluated.

5 subjects may receive elective surgical treatment within the prophylaxis treatment period (after the first drug administration in day 0).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥12 years old and ≤65 years old;
* Male patients who are clinically diagnosed with severe (laboratory tested FVIII:C <1%) hemophilia A, including historical FVIII:C <1%;
* Previously received FVIII treatment (prophylactic or bleeding treatment), have the relevant records and are verified to have accumulated exposures days( EDs) ≥150 days;
* The bleeding treatment records of at least 3 months before screening can be obtained;
* Negative FVIII inhibitor assay results (laboratory tested Nijmegen-Bethesda assay result <0.6 BU(Bethesda unit)/mL);
* The prothrombin time is normal or international normalized ratio (INR) ≤1.5; 7. Platelet count ≥100 × 109/L;

Exclusion Criteria:

* Known allergy to recombinant coagulation factor VIII concentrate or any excipient; known allergy to bovine, rodent or hamster bovine;
* Has a history or family history of blood coagulation factor VIII inhibitor;
* Clinical liver function test (glutamic-pyruvic transaminase, glutamic-pyruvic transaminase) ≥ three times the upper limit of normal (ULN) or clinical kidney function test (blood urea nitrogen, creatinine) ≥ three times the ULN;
* Patients clinically diagnosed with active Hepatitis B or Hepatitis C;
* Patients with other coagulation dysfunction diseases in addition to hemophilia A;
* Patients with severe heart disease, including myocardial infarction and cardiac dysfunction of class III or above;
* Patients who previously experienced intracranial bleeding;

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Hemophilia A is a kind of sex chromosome recessive genetic disease and ofter occurs in male.
Enrollment: 73 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Annualized Bleeding Rate | up to 24 weeks
  Annualized Bleeding Rate（ABR） can be calculated using the following formula: Number of bleeding events in efficacy evaluation period/(number of days in treatment period/365.25)

SECONDARY OUTCOMES:
Annualized joint bleeding rate | up to 24 weeks
  Annualized joint bleeding rate（AJBR） can be calculated using the following formula: Number of joint bleeding events during efficacy evaluation period/(number of days in treatment period/365.25).
FVIII incremental in-vivo recovery | Predose within 30 min，15 min±2 min、1 hour±5 min.
  Incremental recovery is determined as the peak factor level recorded in the first hour after infusion and is reported as [IU/ml]/[IU/kg]
Bleeding event treatment efficacy | up to 24 weeks
  The investigator shall evaluate the hemostatic effect after the treatment of every bleeding event of subjects based on a four-point scale(excellent, good, moderate, not relieved).
Elimination Half Life | Predose within 30 min，15 min±2 min、30 min±2 min，1 hour±5 min，3 hours±5 min，6 hours±5 min，9 hours±10 min，12hours h±10 min，24 hours±10 min，28 hours±10 min，32 hours±10 min and 48 hours±10 min post-dose.
  t1/2; One-stage aPTT Clotting Assay and Chromogenic Assay
Clearance | Predose within 30 min，15 min±2 min、30 min±2 min，1 hour±5 min，3 hours±5 min，6 hours±5 min，9 hours±10 min，12hours h±10 min，24 hours±10 min，28 hours±10 min，32 hours±10 min and 48 hours±10 min post-dose.
  CL; One-stage aPTT Clotting Assay and Chromogenic Assay
Area Under the Curve to the Last Measurable Timepoint | Predose within 30 min，15 min±2 min、30 min±2 min，1 hour±5 min，3 hours±5 min，6 hours±5 min，9 hours±10 min，12hours h±10 min，24 hours±10 min，28 hours±10 min，32 hours±10 min and 48 hours±10 min post-dose.
  AUClast;One-stage aPTT Clotting Assay and Chromogenic Assay

OTHER OUTCOMES:
Incidence of FVIII inhibitors | up tp 24 weeks
  The Nijmegen-Bethesda assay shall be used to monitor the production of FVIII inhibitors during the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Renchi Yang, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin, China